CLINICAL TRIAL: NCT04469270
Title: An Adaptive, Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Engensis in Participants With Painful Diabetic Peripheral Neuropathy
Brief Title: Study to Assess Safety and Efficacy of Engensis in Painful Diabetic Peripheral Neuropathy
Acronym: REGAiN-1A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMDN-003-2
Record Dates: First submitted 2020-06-25; First posted 2020-07-14 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Engensis (Experimental): 16 (ea) 0.25mg (0.5 mL) injections in each of the right and left gastrocnemius muscles on Days 0, 14, 90, and 104.
  Interventions: Biological: Engensis
- Placebo (Placebo Comparator): 16 0.5 mL injections in each of the right and left gastrocnemius muscles on Days 0, 14, 90, and 104.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Engensis — Intramuscular injections
  Arms: Engensis
Other: Placebo — Intramuscular injections
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intramuscular administration of Engensis on pain in participants with painful diabetic peripheral neuropathy in the feet and lower legs, as compared to Placebo, as a second Phase 3, well controlled study, sufficient in supporting the efficacy and safety of Engensis.

DETAILED DESCRIPTION:
Overall Design VMDN-003-2 is an adaptive Phase 3, double-blind, randomized, placebo-controlled, multicenter study designed to assess the efficacy and safety of Engensis (containing the active pharmaceutical ingredient VM202) in Participants with painful Diabetic Peripheral Neuropathy. Following completion of the informed consent process, Screening activities (during 45 days [from Day -52 to Day -7] prior to Day 0) will determine which Participants meet all-but-one eligibility criteria, which are assessed by an adjudication procedure, followed by completion of a 7-day eDiary prior to Day 0. Eligible participants will be enrolled and randomly assigned in a double-blind fashion and in a 1:1 ratio on Day 0 to either Engensis or Placebo. During Screening, medical history and familial cancer history, demographics, vital signs, height, body mass index, waist size, physical examination, retinal fundoscopy (by an ophthalmologist), 12-lead electrocardiogram, ultrasound of the right and left gastrocnemius muscles (to guide Study Injections), laboratory assessments, estimated glomerular filtration rate, Hemoglobin A1c levels, viral screening, a record of all concomitant medications and procedures, urine drug analysis, and urine pregnancy test for females of childbearing potential will be conducted.

In addition, the following procedures will be conducted during Screening: Hospital Anxiety and Depression Scale, Accurate Pain Reporting and Placebo Response Reduction, Michigan Neuropathy Screening Instrument, and cancer screening tests.

During 7 days before Day 0 and randomization, Participants must complete the full Brief Pain Inventory for Diabetic Peripheral Neuropathy on an eDiary for determining the Average Daily Pain Scores for at least 5 out of the 7 days. Adverse event assessments will start upon completion of the consent process at the start of Screening.

At any time prior to dosing on Day 0, Bedside Sensory Testing should be administered.

Following randomization, and prior to the first intramuscular injections of Engensis or Placebo on Day 0, the partial Brief Pain Inventory for Diabetic Peripheral Neuropathy, , and quality of life instruments will be completed. Blood will be collected for testing of selected cytokines, anti-Hepatic growth factor antibodies, and laboratory assessments.

All Participants will receive sixteen (16) 0.5-mL intramuscular injections of Engensis or Placebo in each calf gastrocnemius muscle at each of two Visits during two Treatment Cycles: Treatment Cycle 1 on Day 0 and Day 14, and Treatment Cycle 2 on Day 90 and Day 104. At 2 hours (± 1 hour) after completion of intramuscular injections of Engensis or Placebo on Days 0 and 14 and Days 90 and 104, vital signs and blood draw for cytokine levels will be performed. Treatment-emergent adverse event assessment, including injection site reactions, will start as of randomization (Day 0) and continue throughout the study.

Follow-up Study Visits will be conducted on Days 28, 60, 150, and 180 or early termination. Vital signs will be recorded at all Study Visits. At the Day 180 Visit (end of study), the following assessments will be conducted: the full Brief Pain Inventory for Diabetic Peripheral Neuropathy (performed for 7 days prior to the Day 180 Visit), Michigan Neuropathy Screening Instrument, Bedside Sensory Testing, Patient Global Impression of Change and the quality of life assessments (36-item Short Form Health Survey and European Quality of Life Health Utilities Index, urine drug analysis, retinal fundoscopy, physical examination, concomitant medications and procedures, and anti-Hepatic Growth Factors antibodies. Blood will be drawn for determination of serum chemistry, lipid profile, pregnancy status, hematology, and Hemoglobin A1c levels. The purpose of this study is to assess the efficacy and safety of Engensis compared to Placebo as measured by changes in the means of the Average Daily Pain Scores of the full Brief Pain Inventory for Diabetic Peripheral Neuropathy, selected blood cytokines, Bedside sensory testing, and assessments of injection site reactions, physical examination, laboratory assessments, vital signs, treatment emergent Adverse events, and serious adverse events.

Study and Treatment Duration:

Screening will occur up to 52 days prior to Baseline (Day 0) and Participants will be followed from Day 0, the day of first Study Injections, to Day 180/Early termination.

Visit Frequency: Consented Participants will be seen and evaluated for enrollment during Screening (up to 52 days prior to Baseline, Day 0). There are 8 visits to the Clinical Site during the study from Day 0 to Day 180 for Study Injections and follow-up.

Intervention Groups and Duration:

Two treatment groups of Participants (Engensis or Placebo) will be in the study for 180 days.

Number of Participants (N = 152 to approximately 250):

The target sample size is a minimum of 152 Participants and the maximum sample size is 250 Participants based on the proposed adaptive design analysis. The final sample size of Participants to be enrolled and evaluated will be determined by the independent Data Monitoring Committee. An interim analysis will be conducted after approximately 50% of Participants in the target sample (i.e., 76 Participants) have completed the primary efficacy endpoint at Day 180 or have withdrawn prematurely. The Data monitoring committee will make a recommendation based on an unblinded (comparative) power analysis.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants age ≥ 18 years at time of completion of the informed consent process
2. Type 1 or 2 diabetes mellitus and on current Standards of Medical Care in Diabetes - 2020 optimal guideline-directed medical therapy in participants (including vaccine recommendations if possible), and without unstable diabetes or significant medical problems, such as progressive end-organ disease, within 3 months of or during Screening, in the judgment of the Investigator
3. Glycosylated HbA1c of ≤ 10.0% using the first assessment collected during Screening
4. Documented diagnosis of bilateral painful diabetic peripheral neuropathy in both lower extremities at least 6 months prior to Screening
5. An Average Daily Pain Score ≥ 4 (standard deviation ≥ 0.3 and ≤ 1.5) that was completed during the 7 days prior to randomization (Day 0)
6. The physical examination component of the Michigan Neuropathy Screening Instrument score of ≥ 2.5
7. If on medication for painful diabetic peripheral neuropathy (other than gabapentin or pregabalin), must have been on a stable dose defined as < 50% change in total dose over 3 months prior to completion of informed consent
8. Male participants and their female partners had to agree to use double-barrier contraception during the study or provide proof of postmenopausal state (minimum 1 year) or surgical sterility
9. Male participants were not to donate sperm during the study
10. Female participants had to be nonpregnant, nonlactating, and either postmenopausal for at least 1 year, or surgically sterile for at least 3 months, or agreed to use double-barrier contraception from 28 days prior to randomization and/or their last confirmed menstrual period prior to study randomization (whichever is longer) until the end of the study
11. Capable and willing to comply with the requirements and restrictions of the protocol and informed consent form
12. Able to complete all screening activities within 52 days of signing the informed consent form.

Exclusion Criteria

1. Other sources of pain that prevented accurate assessment of diabetic peripheral neuropathy pain (e.g., thoracic and/or lumbar root proximal neuropathy, mononeuritis multiplex)
2. Peripheral neuropathy caused by a condition other than diabetes: e.g., anatomic (sciatic nerve compression), systemic (monoclonal gammopathy), metabolic (thyroid disease), and toxic (alcohol use) neuropathies
3. Had taken gabapentin or pregabalin during 30 days before completion of informed consent process or was going to take at any time during the study
4. Progressive or degenerative neurological disorder, such as amyotrophic lateral sclerosis, Alzheimer's disease, Parkinson's disease, vascular dementia, multiple sclerosis, or other neurological disorders determined by the Investigator to preclude participation
5. Symptomatic peripheral artery disease or peripheral artery disease requiring revascularization and/or that may interfere with the conduct of the study
6. Vasculitis, such as from Buerger's or other diseases
7. Systolic blood pressure >180 mmHg on tolerable doses of standard antihypertensive medications at Screening determined by the Investigator to preclude participation
8. Hyperlipidemia or dyslipidemia not being treated with an optimal treatment regimen that follows the Standards of Care for hyperlipidemic/dyslipidemic patients with DM
9. Class 3 or 4 heart failure
10. Symptomatic bradycardia or untreated high degree atrioventricular block
11. Stroke or cerebrovascular accident or myocardial infarction within 3 months before Screening
12. Estimated glomerular filtration rate < 30 mL/min/1.73 m2 using the chronic kidney disease epidemiology collaboration formula based on Cystatin C levels
13. Progressive renal dysfunction, defined as a decrease in estimated glomerular filtration rate to chronic kidney disease Stage 1, 2, or 3 in the past 6 months before Screening
14. Ophthalmologic conditions pertinent to signs or symptoms of proliferative diabetic retinopathy or other ocular conditions that precluded standard ophthalmologic examination
15. Myopathy (e.g., Duchenne or Becker muscular dystrophy, polymyositis)
16. Any prior or planned lower extremity amputation (excluding toe amputations) due to diabetic complications or prior lower leg injury (e.g., scarring, muscle atrophy) in the calf area (gastrocnemius) that would significantly reduce the surface area of the skin or amount of intact skeletal muscle required for the 16 treatment injections of Engensis
17. Active infection requiring antimicrobial agent(s) (chronic infection or severe active infection that may compromise the Participant's well-being or participation in the study, in the Investigator's judgment)
18. Chronic inflammatory or autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis)
19. Immunosuppression due to underlying disease (e.g., rheumatoid arthritis, systemic lupus erythematosus) or to currently receiving immunosuppressive drugs, (e.g., chemotherapy, corticosteroids) or to radiation therapy
20. Participants requiring chronic oral or injectable steroids and unwilling to refrain from taking these drugs for the duration of the study
21. Participants with a family medical history of 2 or more first-degree relatives (parent, sibling, child) diagnosed to have the same type of cancer - breast cancer, cervical cancer, colon cancer, endometrial cancer, lung cancer, or prostate cancer; or with a family medical history of Lynch Syndrome (hereditary non-polyposis colorectal cancer) in any first-degree relative; or who show positive results during cancer screening
22. Positive human immunodeficiency virus or human T-cell lymphotropic virus I/II test at Screening
23. Participants with cancer who have not been cancer-free for ≥5 years with the following exceptions (not excluded): Participants with in-situ basal cell or squamous cell carcinoma
24. Participants with a prior history of stem cell transplant for cancer no matter how long they have been cancer-free
25. Active acute or chronic hepatitis B
26. Active hepatitis C
27. Clinically significant laboratory values or current medical conditions during Screening that, in the judgment of the Investigator, should be exclusionary
28. Hospital Anxiety and Depression Scale score of ≥ 15 on either subscale
29. History of drug abuse (the habitual taking of addictive or illegal drugs) in the past 3 months and positive for Drugs of Abuse, with the exception of cannabis, during Screening
30. Participants unwilling to discontinue their use of the following during Screening at least 7 days before starting eDiary entries and not use any of the following during the study:

    * skeletal muscle relaxants
    * opioids
    * transcutaneous electrical nerve stimulation (tens)
    * acupuncture
    * benzodiazepines (other than stable bedtime dose)
    * injectable or oral steroids
31. Participants not on a stable dose and not willing to remain on a stable dose during study for the following drugs:

    * antidepressants
    * antiepileptics
    * duloxetine
32. Participants using the following medications and unwilling to discontinue topical use on the lower legs and feet and throughout the study:

    * capsaicin
    * anesthetic creams (except during Study Injections)
    * anesthetic patches
    * isosorbide dinitrate spray
33. Use of an investigational drug or treatment in past 30 days or previous participation in a clinical study with Engensis
34. Body mass index ≥ 42 kg/m2
35. Recent treatment for COVID-19 with ongoing sequelae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Trials - Little Rock, Little Rock, Arkansas
  - California Medical Clinic for Headache, Los Angeles, California
  - Clinical Trials Research - Sacramento, Sacramento, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Gateway Clinical Trials, LLC, O'Fallon, Illinois
  - Foot & Ankle Center of Illinois, Springfield, Illinois
  - Clinical Research Professionals, Chesterfield, Missouri
  - Richmond Behavioral Associates, Staten Island, New York
  - Health Concepts, Rapid City, South Dakota
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - ClinPoint Trials LLC, Waxahachie, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engensis | Placebo
Started | 81 | 81
Completed (Completed Day 180 visit) | 65 | 75
Not Completed | 16 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Not Dosed - 2 subjects misrandomized, included in ITT, but not Safety population. | 2 | 0
Not completed — missing | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis | Placebo | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 51 | 98
  >=65 years | 34 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.46) | 61.0 (10.25) | 61.8 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 58 | 56 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 69 | 70 | 139
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 162
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.533 (5.2182) | 31.440 (4.7049) | 31.987 (4.9830)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Engensis Compared to Placebo Painful Diabetic Peripheral Neuropathy in Feet and Lower Legs Comparing Average Daily Pain Score From Day 0 Visit to Day 180 Visit on Brief Pain Inventory for Participants With Diabetic Peripheral Neuropathy
Description: • The Brief Pain Inventory for Participants with Diabetic Peripheral Neuropathy has a minimum score of 0 and a maximum score of 10, with a higher score representing a worse outcome of more pain. Change in Baseline to Day 180.
  Summary of the Actual Value of the Change from Baseline to Day 180 in Average Daily Pain Score (Intent-To-Treat Population).
  Overall Engensis n=79.
Time Frame: 180 days
Population: Summary of the Actual Value of the Change from Baseline to Day 180.
  81 subjects were randomized to Engensis. Two Engensis subjects were never dosed and were withdrawn from the study on Day 0, therefore do not fall into the safety population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 79 | 81
score on a scale | -2.03 (2.020) | -2.69 (2.115)

2. Secondary Outcome: Efficacy of Engensis on Worst Pain in Painful Diabetic Peripheral Neuropathy in Feet and Legs by Comparing Change From Baseline (Day 0) in Worst Pain Score From Brief Pain Inventory for Diabetic Peripheral Neuropathy to Day 180 Compared to Placebo
Description: • The Brief Pain Inventory for Diabetic Peripheral Neuropathy has a minimum score of 0 and a maximum score of 10, with a higher score representing a worse outcome of more pain. Summary of the Actual Value of the Change from Baseline to Day 180 in Worst Pain Score (Intent-To-Treat Population).
Time Frame: 180 days
Population: Summary of the Actual Value of the Change from Baseline to Day 180 in Worst Pain Score (Intent-To-Treat Population).
  81 subjects were randomized to Engensis. Two Engensis subjects were never dosed and were withdrawn from the study on Day 0, therefore do not fall into the safety population. Overall Engensis n=79.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 79 | 81
score on a scale | -2.10 (2.374) | -3.06 (2.588)

3. Secondary Outcome: Efficacy of Engensis Reducing Painful Diabetic Peripheral Neuropathy in Feet and Legs by Determining a ≥ 50% Reduction in the Average Daily Pain Score From Baseline to Day 180 Using the Brief Pain Inventory With Participants Diabetic Peripheral Neuropathy
Description: • The Average Daily Pain Score from the Brief Pain Inventory for Participants with Diabetic Peripheral Neuropathy has a minimum score of 0 and a maximum score of 10 with a higher score representing a worse outcome of more pain. Summary of Responders with ≥50% Reduction from Baseline in the Average Daily Pain Score on Day 180 (Intent-To-Treat Population).
Time Frame: 180 days
Population: Responders with ≥50% Reduction from Baseline in the Average Daily Pain Score on Day 180 (Intent-To-Treat Population).
  81 subjects were randomized to Engensis. Two Engensis subjects were never dosed and were withdrawn from the study on Day 0, therefore do not fall into the safety population. Overall Engensis n=79.
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 79 | 81
Participants | 24 | 33

4. Secondary Outcome: Safety of Engensis in Painful Diabetic Peripheral Neuropathy in Feet and Legs Comparing Incidence of Adverse and Serious Adverse Events, Incidence of Injection Site Reactions, and Incidence of Clinically Significant Laboratory Values to Placebo
Description: To evaluate the safety of intramuscular administration of Engensis in Participants with painful diabetic peripheral neuropathy in the feet and lower legs as compared to Placebo.
  • Incidence of adverse events and serious adverse event; Incidence of injection site reactions; Incidence of clinically significant laboratory values.
Time Frame: 180 days
Population: Overall Summary of Incidence of Treatment-Emergent Adverse Events (Safety Population) by Severity, Incidence of Injection Site Reactions, and Incidence of Clinically Significant Laboratory Values.
  81 subjects were randomized to Engensis, Two Engensis subjects were never dosed and were withdrawn from the study on Day 0, therefore do not fall into the safety population. Overall Engensis n = 79.
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 79 | 81
Participants
  Any Treatment Emergent AE | 45 | 44
  Treatment Emergent AE by Severity - Mild | 18 | 24
  Treatment Emergent AE by Severity - Moderate | 20 | 17
  Treatment Emergent AE by Severity - Severe | 7 | 3
  Injection Site Reactions | 10 | 9
  Clinically Significant Lab Values - Any Abnormal Analyte Value of Interest | 29 | 30

5. Secondary Outcome: To Evaluate the Possibility of Cellular Responses to Engensis
Description: Change from baseline in the TNF-alpha, IL-1b, IFNy, IL-6, IL-4, IL-10, and IL-12p70 cytokine profile post-dose at the Day 104 visit.
Time Frame: 104 days
Population: Change from baseline in the TNF-alpha, IL-1b, IFNy, IL-6, IL-4, IL-10, and IL-12 p70 cytokine profile post-dose at the Day 104 visit.
  Of the 79 Engensis Subjects that were dosed, 69 had Cytokine Samples collected at both Day 0 and Day 104. Of the 81 Placebo Subjects that were dosed, 77 had Cytokine Samples collected at both Day 0 and Day 104.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 69 | 77
ng/L
  TNF-alpha - Change from Baseline Day 104 | -0.334 (4.5971) | 0.518 (1.8213)
  IL-1beta - Change from Baseline Day 104 | -0.245 (2.0345) | -0.001 (0.0125)
  IF-gamma - Change from Baseline Day 104 | -3.371 (27.8190) | 1.087 (5.4897)
  IL-6 - Change from Baseline Day 104 | -0.262 (1.6692) | 0.012 (0.6282)
  IL-4 - Change from Baseline Day 104 | -0.002 (0.0157) | 0.0 (0.0)
  IL-10 - Change from Baseline Day 104 | 0.147 (1.2292) | 0.029 (0.1439)
  IL-12 - Change from Baseline Day 104 | 0.0 (0.0) | 0.0 (0.0)

6. Secondary Outcome: To Evaluate the Possibility of Humoral Responses to Engensis - Anti-Hepatic Growth Factor
Description: • Presence of anti-hepatocyte growth factor antibodies following Engensis administration compared to Placebo
  - Anti-hepatocyte growth factor antibodies will be collected on Day 0, 60, 90, 150 and 180, and the presence will be summarized according to each time point.
Time Frame: Days 0, 60, 90, 150 and 180
Population: Safety Population. 81 subjects were randomized to Engensis. Two Engensis subjects were never dosed and were withdrawn from the study on Day 0, therefore do not fall into the safety population. Overall Engensis n=79.
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 79 | 81
Participants
  Day 0 - Anti-HGF Present | 0 | 0
  Day 60 - Anti-HGF Present | 0 | 0
  Day 90 - AntiHGF Present | 1 | 0
  Day 150 - AntiHGF Present | 0 | 1
  Day 180 - AntiHGF Present | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) to Day 180
Description: Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Safety Populations
Arm/Group | Engensis | Placebo
All-Cause Mortality (participants affected / at risk) | 1/79 | 0/81
Serious Adverse Events (participants affected / at risk) | 7/79 | 4/81
Other Adverse Events (participants affected / at risk) | 38/79 | 41/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=79) | Placebo (N=81)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=79) | Placebo (N=81)
COVID-19 (Infections and infestations) | 4 (4) | 4 (4)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 4 (4)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Macular oedema (Eye disorders) | 1 (1) | 1 (1)
Retinal haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergenic (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Retinal scar (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 4 (4) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (Infections and infestations) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site scar (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Electric shock sensation (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophasphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Plueral effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study is part of a multi-center research study, and publication of the results of the Study conducted at the Site shall not be made before the first multi-center publication by Sponsor. If there is not a multi-center publication within eighteen (18) months after the Study has been completed or terminated at all Study sites, and all data has been received, Site shall have the right to publish its results from the Study, subject to the following notice requirements.

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04469270/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04469270/SAP_001.pdf